CLINICAL TRIAL: NCT06016803
Title: Evaluation of the Tolerance of the Medical Device RL3010A - DP0378 in Children and Adults Presenting a Superficial Wound After a Dermatological Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RL3010A2022001
Record Dates: First submitted 2023-07-25; First posted 2023-08-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Skin Abrasion; Superficial Wound
Keywords: Wound healing; Medical device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Subjects having undergone a Cryotherapy for benign cutaneous lesions, warts, or hyperpigmentation (Experimental): Group applying the tested medical device
  Interventions: Device: Cicatryl (RL3010A - DP0378)
- Subjects having undergone a Laser or IPL procedure for dermatological or aesthetical indications (Experimental): Group applying the tested medical device
  Interventions: Device: Cicatryl (RL3010A - DP0378)
- Subjects having undergone a skin lesion excision for which stitches were removed (Experimental): Group applying the tested medical device
  Interventions: Device: Cicatryl (RL3010A - DP0378)

INTERVENTIONS:
Device: Cicatryl (RL3010A - DP0378) — Tested product is applied twice a day. The maximum duration of application is 7 days.

SUMMARY:
The CE-marketed medical device class IIa RL3010A - DP0378 developed by Pierre Fabre Laboratories is indicated in the treatment of superficial wounds and abrasions. It forms a protective layer on the surface of wounds maintaining a moist environment improving the healing process thanks to its moisturizing and film-forming effect.

Through this study, the overall tolerance of the medical device will be evaluated in subjects presenting a superficial wound after having undergone a dermatological procedure as cryotherapy, laser (laser Nd Yag, fractional laser C02), Intense Pulse Light (IPL) or skin lesion excision for which stitches were removed.

DETAILED DESCRIPTION:
This open-labelled study will be conducted as a monocentric study, in children and adults presenting a superficial wound after having undergone a dermatological act.

To assess the global tolerance of the medical device RL3010A - DP0378 in subjects presenting a superficial wound after having undergone a dermatological procedure, after 7 days of twice daily applications under normal conditions of use

3 visits are planned:

* Visit 1: Inclusion (D1)
* Visit 2: Intermediate visit (D3)
* Visit 3: Final visit (D8)

The maximal duration of participation for a subject is 8 days, from the inclusion visit (visit 1) to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject who just undergone (the same day) a dermatological procedure, done according to the investigator's usual practices:

  * Group 1: Cryotherapy for benign cutaneous lesions, warts, or hyperpigmentation
  * Group 2: Laser (laser Nd Yag, fractional laser C02) or Intense pulse Light (IPL) procedure for dermatological or aesthetical indications (including tattoo removal and depilation)
  * Group 3: Skin lesion excision for which stitches were removed
* Subject with a superficial wound after the dermatological procedure

Exclusion Criteria:

Criteria related to the skin condition :

* Subject having received artificial UV exposure, excessive or prolonged exposure to natural sunlight on the studied area within 4 weeks before the inclusion visit or planning to be exposed to artificial UV, excessive or prolonged natural sunlight during the study
* Subject having a skin disease, skin abnormalities, or dermatological condition on the studied area other than the indication of the dermatological procedure liable to interfere with the study assessments (including infectious or inflammatory dermatosis, photodermatosis, etc.)
* Subject with a known history of allergy or contact dermatitis caused by any of the ingredients of the tested product, antiseptic, dressing or latex (if used by the center)
* Subject with healing disorders
* Subject with coagulation disorders
* Knowledge of Acquired Immunodeficiency Syndrome or Infectious (acute) Hepatitis
* Other acute, chronic or progressive disease or medical history considered by the investigator hazardous for the subject or incompatible with the study or liable to interfere with the study assessments

Criteria related to treatments and/or products :

* Systemic corticosteroid treatment in the 4 weeks prior to the inclusion visit or ongoing or planned to be started during the study
* Systemic antibiotics treatment in the 2 weeks prior to the inclusion visit, ongoing or planned to be started during the study
* Systemic treatments that may affects homeostasis (anticoagulant therapy, platelet aggregation inhibitor) in the 4 weeks prior to the inclusion visit, ongoing or planned to be started during the study
* Any other systemic treatment that may affect the healing process, or incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study
* Topical steroid, non-steroid anti-inflammatory, immunomodulator and antibiotics treatments applied on the tested area in the 2 weeks prior to the inclusion visit, ongoing or planned to be started during the study
* Any topical repairing treatment or product applied on the tested area between the dermatological procedure (stitch removal for group 3) and the inclusion visit
* Any other topical treatment on the tested area that may affect the healing process, or incompatible with the study or liable to interfere with the study assessments according to the investigator, in the weeks prior to the inclusion visit, ongoing or planned to be started during the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
To assess the global tolerance of the medical device RL3010A - DP0378 in subjects presenting a superficial wound after having undergone a dermatological procedure, after 7 days of twice daily applications under normal conditions of use | Day 8
  Global tolerance with 5 levels ranked from best to worst : Excellent (No functional nor physical signs related to the investigational product observed or reported by the subjects) - Very good - Good - Moderate - Bad

SECONDARY OUTCOMES:
To assess the evolution of the physical signs of local tolerance at the site of product application on the wound | Day 1 before and immediately after the test product application (10 to 30 minutes), at Day 3 and at Day 8.
  Physical signs with 5 levels ranked from best to worst : None - Very mild - Mild - Moderate - Severe
To assess the evolution of the functional signs of local tolerance at the site of product application on the wound | Day 1 before and immediately after the test product application (10 to 30 minutes), at Day 3 and at Day 8.
  Functional signs with 5 levels ranked from best to worst : None - Very mild - Mild - Moderate - Severe
To assess the repairing efficacy of the product | Day 3 and Day 8
  Scale with 4 levels ranked from worst to best : Not effective - Little effective - Effective - Very effective
To assess the soothing efficacy of the product | Day 3 and Day 8
  Scale with 4 levels ranked from worst to best : Not effective - Little effective - Effective - Very effective
To assess the soothing efficacy of the product | Day 1 before and immediately after the test product application, at Day 3 and at Day 8
  Discomfort sensations with NRS ranging from 0 (None) to 10 (Hugely). Higher scores mean a worse outcome.
To evaluate subjects' global satisfaction as regards to the use the medical device RL3010A - DP0378. | Day 3 and Day 8
  Global satisfaction through a specific questionnaire (Conditions of use, organoleptic properties, effects, and others will be assessed).
To evaluate the compliance of the subjects to product application. | About 8 days
  The subject / subject's parent(s) will report in his/her diary the applications of investigational product and any omissions or changes in the frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermscan Poland, Gdansk, Poland, Poland